CLINICAL TRIAL: NCT01350154
Title: Does Modulation of the nNOS System in Patients With Muscular Dystrophy and Defect nNOS Signalling Affect Cardiac, Muscular or Cognitive Function?
Brief Title: Effect of Modulating the nNOS System on Cardiac, Muscular and Cognitive Function in Becker Muscular Dystrophy Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Christina Kruuse, Senior Registrar, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RHGLBMD
Record Dates: First submitted 2011-05-04; First posted 2011-05-09 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Becker Muscular Dystrophy
Keywords: clinical trial; sildenafil; revatio; muscular dystrophy; adult; nNOS
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophies | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sildenafil (Revation) 20 mg (Experimental): This arm will receive sildenafil for 4 weeks followed by 2 weeks washout and 4 weeks placebo.
  Interventions: Drug: Sildenafil
- Placebo (Experimental): This arm will receive placebo for 4 weeks followed by 2 weeks washout and 4 weeks sildenafil
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sildenafil — 20 mg in gelatine capsules, oral, three times daily
  Other Names: Placebo
  Arms: Sildenafil (Revation) 20 mg
Drug: Placebo — Lactose monohydrate oral in gelatine capsules, 3 times daily
  Other Names: Sildenafil (Revatio)
  Arms: Placebo

SUMMARY:
This study is done to evaluate whether treatment with the drug sildenafil (Revatio®) can improve muscular, cardiac, cerebrovascular or cognitive function in patients with Beckers muscular dystrophy when compared to placebo (inactive medication). The study is based on the recent findings of an improved cardiac function in a mouse model of muscular dystrophy (Adamo et al 2010) and the previous findings of changed cognitive function in people with Becker dystrophy.

In muscular dystrophy, the cellular protein, dystrophin is affected. During normal conditions, the enzyme neuronal nitric oxide synthase (nNOS), which produce nitric oxide (NO), is attached to dystrophin. NO is important in normal vascular function in each of muscle, heart and brain by stimulating production of cyclic GMP. However, in muscular dystrophy with dystrophin deficiency, nNOS do not have the normal cellular anchor, resulting in decreased NO levels and subsequent reduced cyclic GMP production. Sildenafil inhibits degradation of cGMP thus prolonging and increasing a cGMP response. Such effects are the basis for use of sildenafil in pulmonary hypertension and erectile dysfunction. Current hypothesis: Sildenafil restores the cyclic GMP function affected in muscular dystrophy wit nNOS deficiency resulting in improved muscle, cardiac, cerebrovascular and cognitive function.

DETAILED DESCRIPTION:
The current clinical trial including people with Becker's muscular dystrophy and established deficiency in muscular content of nNOS protein consist of three sub-studies focusing on each of muscle function, cardiac function and brain function. In muscular dystrophy the dystrophin cellular complex usually located to muscle cells, is disrupted resulting in a known reduced nNOS activity. The reduced nNOS leads to reduced cyclic GMP production. nNOS and cyclic GMP are involved in the vascular response in striate muscle, cardiac vessels as well as the cerebrovascular response to hypercapnia and regional activation. In muscular dystrophy, the is an affected muscular and cardiac function and in some patients a changed cognitive function in described. Whether such is related to a reduced nNOS function and subsequent cGMP production is not fully understood. Inhibition of cGMP degradation by inhibiting the cGMP degrading enzyme phosphodiesterase 5 (PDE5) using PDE5 inhibitors such as sildenafil may result in restoration of vascular responses.

The study is designed as a double blind, randomised, balanced, placebo-controlled cross-over study performed during a 10 week treatment period. The patients will receive 4 weeks of either sildenafil or placebo with a 2 week washout period in between treatments. The study out-come parameters will be performed on two consecutive days at baseline, 4 weeks and 10 weeks, at two collaborating centers, Rigshospitalet for muscle and cardiac parameters and Glostrup Hospital for cerebrovascular and cognitive parameters.

The primary endpoints relate to each sub-study, assessing and comparing individual changes from baseline and during placebo/sildenafil treatment.

ELIGIBILITY:
Inclusion Criteria:

* Muscular dystrophy with known deficiency in nNOS
* Reduced cardiac function (<50%) and/or reduced muscular function (MRC<4+)
* Stable dosing (> 3 month)of cardiovascular medication
* Signed informed consent

Exclusion Criteria:

* Recent (< 6 month) cerebral or cardiac stroke
* Use of nitrate containing compounds, alpha receptor blocking agents or potent CUP3A4 inhibitors.
* Intolerance or allergy to sildenafil, or intake of drugs not compatible with sildenafil intake
* Overuse of drugs or alcohol
* inclusion in other trials of experimental medication within last 30 days
* known epilepsy
* reduced liver function (ASAT >500U/l in 2 repeated measurements when corrected for increase in creatinkinase levels.
* non-arteriitis anterior ischemic optic neuropathy (NAION) with reduced vision
* contraindications for MRI scan (metal implants, claustrophobia)
* hypotension (<90 mmHg systolic at baseline)
* conditions, medical or psychosocial which makes the subject inclusion inadvisable

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-11; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Difference in change from baseline to 4 week placebo/sildenafil treatment in handgrip test with concomitant ultrasound measurement of flow in the brachial artery | Baseline and 4 weeks treatment
  Primary outcome for substudy 1
Difference in changes from baseline to 4 week placebo/sildenafil treatment in resting cardiac end-diastolic volume measured by MRI | Baseline and 4 week treatment
  Primary outcome for substudy 2
Difference in changes from baseline to 4 week placebo/sildenafil treatment in cerebrovascular reactivity to CO2 inhalation and finger stimulation measured by BOLD fMRI | Baseline and 4 weeks treatment
  Primary outcome for substudy 3
Difference in changes from baseline to 4 weeks placebo/sildenafil treatment in Cognitive function measured by Cambridge Neuropsychological Test Automated Battery (CANTAB) | Baseline and 4 weeks treatment
  Primay outcome for substudy 3

SECONDARY OUTCOMES:
Difference in changes from baseline to 4 weeks placebo/sildenafil treatment in 6 minutes walk test | Baseline and 4 weeks treatment
  Substudy 1
Difference in changes from baseline to 4 weeks placebo/sildenafil treatment in max test, measured by O2 uptake during maximal exercise on bike | Baseline and 4 weeks treatment
  Substudy 1
Difference in changes from baseline to 4 weeks placebo/sildenafil treatment in Quality of life by SF36 | Baseline and 4 weeks treatment
  Substudy 1
Difference in changes from baseline to 4 weeks placebo/sildenafil treatment in resting cardiac function measured by cardiac MRI | Baseline and 4 weeks treatment
  Substudy 2. Evaluation of resting cardiac ejection fraction and end-systolic volume.
Difference in changes from baseline to 4 weeks placebo/sildenafil treatment in cardiac function during hand grip exercise measured by cardiac MRI | Baseline and 4 weeks treatment
  Substudy 2. Cardiac volumes and ejection fraction during 1 minute repeated maximal force hand exercise will be measured.
Difference in changes from baseline to 4 weeks placebo/sildenafil treatment in cerebrovascular reactivity and blood flow | Baseline and 4 weeks treatment
  Substudy 3. fMRI BOLD evaluation of visual stimulation, MRI angiography for arterial diameter, arterial spin labeling for evaluation of cerebral blood flow and blood volumen.
Difference in changes from baseline to 4 weeks placebo/sildenafil treatment in basic activity and metabolites of the brain | Baseline and 4 weeks treatment
  Substudy 3.Resting state network by fMRI and metabolites in brain regions by MRI spectroskopy.
Difference in changes from baseline to 4 weeks placebo/sildenafil treatment in cognitive function measured by paper and pen test battery | Baseline and 4 weeks treatment
  Substudy 3. A paper and pen cognitive test battery will be applied, including Trail making A and B, Addenbrooke's Cognitive Examination, Symbol DIgital MOdality tests
Difference in changes from baseline to 4 weeks treatment placebo/sildenafil in plasma levels of signalling molecules | Baseline and 4 weeks treatment
  Substudy 3. From blood samples taken at baseline, 4 and 10 weeks, analysis of several signalling molecules relevant for cardiac and cerebrovascular function will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: John Vissing, MD, DMSci, Study Chair — Neuromuscular Clinic and Research Unit, Dept. Neurology, Rigshospitalet
Locations (1):
- Neuromuscular Clinic and Research Unit, Dept. Neurology, Rigshospitalet,, Copenhagen, Denmark